CLINICAL TRIAL: NCT04142242
Title: Safety and Immunogenicity of a Single Dose of MenACYW Conjugate Vaccine at Least 3 Years Following Initial Vaccination With Either Menomune® Vaccine or MenACYW Conjugate Vaccine in Older Adults
Brief Title: Study to Assess the Safety and Immunogenicity of a Single Dose of a Quadrivalent Meningococcal (MenACYW) Conjugate Vaccine in Older Adults Who Received a Primary Vaccination (3 or More Years Earlier) in Study MET49
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MEQ00066; U1111-1217-2058 (Other: UTN)
Record Dates: First submitted 2019-10-24; First posted 2019-10-29 (Actual); Results first posted 2021-04-26 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Meningococcal Infection (Healthy Volunteers)
MeSH Terms: conditions — Meningococcal Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Group 1: MenACYW Conjugate Vaccine (MET 49 - Menomune-primed Participants) (Experimental): Participants who received a single dose of Menomune vaccine in a previous study MET49, provided a blood sample for assessment of antibody persistence (at enrollment [Day 0]) followed by a single intramuscular (IM) dose of MenACYW Conjugate vaccine, at Day 0, during Stage I in the present study (MEQ00066).
  Interventions: Biological: Meningococcal Polysaccharide (serogroups A, C, Y, and W) Tetanus Toxoid Conjugate Vaccine
- Group 2: MenACYW Conjugate Vaccine (MET49 - MenACYW Conjugate Vaccine-primed Participants) (Experimental): Participants who received a single dose of MenACYW Conjugate vaccine in a previous study MET49, provided a blood sample for assessment of antibody persistence (at enrollment [Day 0]) followed by a single IM dose of MenACYW Conjugate vaccine at Day 0, during Stage I in the present study (MEQ00066).
  Interventions: Biological: Meningococcal Polysaccharide (serogroups A, C, Y, and W) Tetanus Toxoid Conjugate Vaccine
- Group 3: MenACYW Conjugate Vaccine (MET49: Menomune-primed Participants) (Experimental): Participants who received a single dose of Menomune vaccine in a previous study MET49, provided a blood sample for assessment of antibody persistence at enrollment (Day 0) during Stage I in the present study (MEQ00066), followed by receiving a single IM dose of MenACYW Conjugate vaccine at Stage II in the present study (MEQ00066).
  Interventions: Biological: Meningococcal Polysaccharide (serogroups A, C, Y, and W) Tetanus Toxoid Conjugate Vaccine
- Group 4: MenACYW Conjugate Vaccine (MET49: MenACYW-primed Participants) (Experimental): Participants who received a single dose of MenACYW Conjugate vaccine in a previous study MET49, provided a blood sample for assessment of antibody persistence at enrollment (Day 0) during Stage I in the present study (MEQ00066), followed by receiving a single IM dose of MenACYW Conjugate vaccine at Stage II in the present study (MEQ00066).
  Interventions: Biological: Meningococcal Polysaccharide (serogroups A, C, Y, and W) Tetanus Toxoid Conjugate Vaccine
- Group 5: Menomune-primed Participants (MET44) (Other): Participants who received a single dose of Menomune vaccine in a previous study MET44, provided a blood sample for assessment of antibody persistence at enrollment (Day 0) during Stage I in the present study (MEQ00066). These participants did not receive any vaccination in the present study (MEQ00066).
  Interventions: Other: Blood sample
- Group 6: MenACYW Conjugate Vaccine-primed Participants (MET44) (Other): Participants who received a single dose of MenACYW Conjugate vaccine in a previous study MET44, provided a blood sample for assessment of antibody persistence at enrollment (Day 0) during Stage I in the present study (MEQ00066). These participants did not receive any vaccination in the present study (MEQ00066).
  Interventions: Other: Blood sample

INTERVENTIONS:
Biological: Meningococcal Polysaccharide (serogroups A, C, Y, and W) Tetanus Toxoid Conjugate Vaccine — Pharmaceutical form: Solution for injection; Route of administration: Intramuscular
  Other Names: MenACYW Conjugate vaccine; MenQuadfi
  Arms: Group 1: MenACYW Conjugate Vaccine (MET 49 - Menomune-primed Participants); Group 2: MenACYW Conjugate Vaccine (MET49 - MenACYW Conjugate Vaccine-primed Participants); Group 3: MenACYW Conjugate Vaccine (MET49: Menomune-primed Participants); Group 4: MenACYW Conjugate Vaccine (MET49: MenACYW-primed Participants)
Other: Blood sample — Blood sample for assessment of antibody persistence.
  Arms: Group 5: Menomune-primed Participants (MET44); Group 6: MenACYW Conjugate Vaccine-primed Participants (MET44)

SUMMARY:
Primary Objective:

To demonstrate sufficiency of the vaccine seroresponse to meningococcal serogroups A, C, W, and Y following administration of a single dose of Meningococcal Polysaccharide (Serogroups A, C, Y, and W 135) Tetanus Toxoid (MenACYW) Conjugate vaccine to Group 1 participants (who received primary vaccination with Menomune vaccine greater than or equal to [>= 3] years earlier at >= 56 years of age in Study MET49).

Secondary Objectives:

Secondary Objective 1 - To demonstrate sufficiency of the vaccine seroresponse to meningococcal serogroups A, C, W, and Y following administration of a single dose of MenACYW Conjugate vaccine to Group 2 participants (who received primary vaccination with MenACYW Conjugate vaccine >= 3 years earlier at >= 56 years of age in Study MET49).

Secondary Objective 2 - To describe vaccine seroresponse rates with respect to serogroups A, C, W, and Y in serum specimens collected 6 days (window, 5-7) post-vaccination in approximately 60 participants from Group 1 (Menomune-primed) and approximately 60 participants from Group 2 (MenACYW Conjugate vaccine-primed).

Secondary Objective 3 - To describe antibody persistence >= 3 years after primary vaccination with Menomune vaccine or MenACYW Conjugate vaccine for participants from all groups.

DETAILED DESCRIPTION:
Study duration per participant in Group 1 and Group 2 was approximately 30 days including: 1 day of screening and vaccination, a phone call and a safety-follow up/end of study visit at Day 8 and Day 30 after vaccine administration, respectively.

Study duration per participant in Group 3 and 4 was approximately 2 years and 30 days including: 1 day of screening, 1 day of vaccination 2 years later, a phone call and a safety-follow up/end of study visit at Day 8 and Day 30 after vaccine administration, respectively.

Study duration per participant in Group 5 and 6 was 1 day.

Safety assessment includes solicited reactions within 7 days after vaccination, unsolicited adverse events (AEs), serious adverse events (SAEs) and adverse event of special interest (AESI)s throughout the study "active phase" (i.e., period of time from revaccination with MenACYW Conjugate vaccine to the end of the short-term [i.e., ~30 days] follow-up after the vaccination).

ELIGIBILITY:
Inclusion criteria:

* Received primary vaccination in Study MET49 or Study MET44 at >= 56 years of age with either Menomune vaccine or MenACYW Conjugate vaccine, as assigned by randomization. (">= 56 years" means from the day of the 56th birthday onwards).
* Able to attend all scheduled visits and to comply with all study procedures.

Exclusion criteria:

* Pregnant, or lactating, or of childbearing potential and not using an effective method of contraception or abstinence from at least 4 weeks prior to vaccination and until at least 4 weeks after vaccination. To be considered of non-childbearing potential, a female must be post-menopausal for at least 1 year, or surgically sterile.
* Participation in the 4 weeks preceding study enrollment/vaccination or planned participation during the active phase of the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure.

Note: "Active phase" refers to the period of time from revaccination with MenACYW Conjugate vaccine to the end of the short-term (i.e., ~30 days) follow-up after the vaccination. Accordingly, following the blood draw at Visit 1, participants in Group 3 and Group 4 will have a 2-year inactive phase prior to Visit 2. Prior to Visit 2, participants in Group 3 and Group 4 will have inclusion and exclusion criteria reassessed and will continue with or be excluded from further participation in the trial as appropriate.

* Receipt of any vaccine in the 4 weeks (28 days) preceding the study vaccination or planned receipt of any vaccine during the active phase of the present study except for influenza vaccination, which might be received at least 2 weeks before or after study vaccine. This exception includes monovalent pandemic influenza vaccines and multivalent influenza vaccines.
* Receipt or planned receipt of any meningococcal vaccine since receipt of a single dose of MenACYW Conjugate vaccine or Menomune vaccine in Study MET49 or Study MET44.
* Receipt of immune globulins, blood, or blood-derived products in the 3 months prior to either enrollment or MenACYW Conjugate vaccination in the current study.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months prior either to enrollment or MenACYW conjugate vaccination in the current study).
* History of meningococcal infection, confirmed either clinically, serologically, or microbiologically.
* At high risk for meningococcal infection during the study (specifically, but not limited to, participants with persistent complement deficiency, with anatomic or functional asplenia, or participants travelling to countries with high endemic or epidemic disease).
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine used in the study or to a vaccine containing any of the same substances (excluding participants in Group 5 and Group 6).
* Verbal report of thrombocytopenia, contraindicating IM vaccination, in the Investigator's opinion (excluding participants in Group 5 and Group 6).
* Personal history of Guillain-Barré Syndrome (GBS) (excluding participants in Group 5 and Group 6).
* Personal history of an Arthus-like reaction after vaccination with a tetanus toxoid-containing vaccine within at least 10 years of the proposed study vaccination (excluding participants in Group 5 and Group 6).
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion (excluding participants in Group 5 and Group 6), contraindicating IM vaccination in the Investigator's opinion.
* Current alcohol abuse or drug addiction.
* Chronic illness that, in the opinion of the Investigator, was at a stage where it might interfere with study conduct or completion.
* Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (temperature >= 100.4°F). A prospective participant should not be included in the study or receive study vaccination until the condition has resolved or the febrile event has subsided.
* Receipt of oral or injectable antibiotic therapy within 72 hours prior to the first blood draw.
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 471 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2022-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (34):
- United States (33):
  - Investigational Site Number 8400026, Chandler, Arizona
  - Investigational Site Number 8400003, San Diego, California
  - Investigational Site Number 8400028, Waterbury, Connecticut
  - Investigational Site Number 8400038, Clearwater, Florida
  - Investigational Site Number 8400023, DeLand, Florida
  - Investigational Site Number 8400007, Jacksonville, Florida
  - Investigational Site Number 8400015, Jacksonville, Florida
  - Investigational Site Number 8400022, Ponte Vedra, Florida
  - Investigational Site Number 8400032, Port Orange, Florida
  - Investigational Site Number 8400020, West Palm Beach, Florida
  - Investigational Site Number 8400027, Newton, Kansas
  - Investigational Site Number 8400017, Wichita, Kansas
  - Investigational Site Number 8400016, Metairie, Louisiana
  - Investigational Site Number 8400010, Elkridge, Maryland
  - Investigational Site Number 8400031, Richfield, Minnesota
  - Investigational Site Number 8400030, St Louis, Missouri
  - Investigational Site Number 8400019, Endwell, New York
  - Investigational Site Number 8400021, Greensboro, North Carolina
  - Investigational Site Number 8400012, Raleigh, North Carolina
  - Investigational Site Number 8400033, Winston-Salem, North Carolina
  - Investigational Site Number 8400013, Fargo, North Dakota
  - Investigational Site Number 8400035, Cincinnati, Ohio
  - Investigational Site Number 8400005, Cincinnati, Ohio
  - Investigational Site Number 8400011, Columbus, Ohio
  - Investigational Site Number 8400014, Uniontown, Pennsylvania
  - Investigational Site Number 8400018, Anderson, South Carolina
  - Investigational Site Number 8400034, Mt. Pleasant, South Carolina
  - Investigational Site Number 8400036, Mt. Pleasant, South Carolina
  - Investigational Site Number 8400024, Dallas, Texas
  - Investigational Site Number 8400001, Murray, Utah
  - Investigational Site Number 8400002, Salt Lake City, Utah
  - Investigational Site Number 8400025, West Jordan, Utah
  - Investigational Site Number 8400004, Charlottesville, Virginia
- Investigational Site Number 6300001, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Robertson CA, Jacqmein J, Selmani A, Galarza K, Oster P. Immune persistence and booster response of a quadrivalent meningococcal conjugate vaccine (MenACYW-TT) 5 years after primary vaccination of adults at >/=56 years of age. Hum Vaccin Immunother. 2024 Dec 31;20(1):2426868. doi: 10.1080/21645515.2024.2426868. Epub 2024 Nov 18. PMID 39555800
- [Derived] Robertson CA, Jacqmein J, Selmani A, Galarza K, Oster P. Immunogenicity and safety of a quadrivalent meningococcal conjugate vaccine (MenACYW-TT) administered as a booster to adults aged >/=59 years: A phase III randomized study. Hum Vaccin Immunother. 2023 Dec 31;19(1):2160600. doi: 10.1080/21645515.2022.2160600. Epub 2023 Jan 11. PMID 36632042
- See also: MEQ00066 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25310&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 04-October-2019 to 02-March-2020 at 34 sites in the United States. A total of 471 participants who received Menomune vaccine or Meningococcal Polysaccharide (Serogroups A, C, Y, and W 135) Tetanus Toxoid (MenACYW) Conjugate vaccine in Study MET49 (NCT02842866) or Study MET44 (NCT01732627) were enrolled and randomized/assigned to a study group in the present study (MEQ00066).
Pre-assignment Details: Study consisted of two stages: Stage I and Stage II. In Stage I, Groups 1 and 2 participants alone received vaccination and Groups 3 and 4 received no vaccination and only provided blood sample for antibody persistence. Groups 3 and 4 participants continued into Stage II and received vaccination in Stage II of the current study.
Period: Stage I
Arm/Group | Group 1: MenACYW Conjugate Vaccine (MET 49 - Menomune-primed Participants) | Group 2: MenACYW Conjugate Vaccine (MET49 - MenACYW Conjugate Vaccine-primed Participants) | Group 3: MenACYW Conjugate Vaccine (MET49: Menomune-primed Participants) | Group 4: MenACYW Conjugate Vaccine (MET49: MenACYW-primed Participants) | Group 5: Menomune-primed Participants (MET44) | Group 6: MenACYW Conjugate Vaccine-primed Participants (MET44)
Started | 139 | 176 | 31 | 39 | 26 | 60
Vaccinated | 138 | 175 | 0 | 0 | 0 | 0
Stage I Full Analysis Set (FAS) (Participants who had a valid serology result for at least 1 serogroup from a pre-vaccination blood sample.) | 138 | 175 | 31 | 39 | 26 | 59
Safety Analysis Set (SafAS) (Participants of Groups 1 and 2 who had received study MEQ00066 vaccine and had available safety data, were analyzed according to the actually received vaccine.) | 151 (1 MenACYW Conjugate vaccine-primed participant was erroneously assigned by Investigator to Group 1 but per planned analysis was counted in Group 2 for safety analysis.) | 162 (14 Menomune-primed participants were erroneously assigned by Investigator to Group 2 but per planned analysis they were counted in Group 1 for safety analysis.) | 0 | 0 | 0 | 0
Completed | 138 | 175 | 31 | 39 | 26 | 59
Not Completed | 1 | 1 | 0 | 0 | 0 | 1
Not completed — Non-compliance with the protocol | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Voluntary withdrawal not due to an adverse event (AE) | 0 | 1 | 0 | 0 | 0 | 0
Period: Stage II
Arm/Group | Group 1: MenACYW Conjugate Vaccine (MET 49 - Menomune-primed Participants) | Group 2: MenACYW Conjugate Vaccine (MET49 - MenACYW Conjugate Vaccine-primed Participants) | Group 3: MenACYW Conjugate Vaccine (MET49: Menomune-primed Participants) | Group 4: MenACYW Conjugate Vaccine (MET49: MenACYW-primed Participants) | Group 5: Menomune-primed Participants (MET44) | Group 6: MenACYW Conjugate Vaccine-primed Participants (MET44)
Started | 0 (Only participants from Group 3 and 4 continued and received vaccination in Stage II part of the study.) | 0 (Only participants from Group 3 and 4 continued and received vaccination in Stage II part of the study.) | 31 | 39 | 0 (Only participants from Group 3 and 4 continued and received vaccination in Stage II part of the study.) | 0 (Only participants from Group 3 and 4 continued and received vaccination in Stage II part of the study.)
Vaccinated | 0 | 0 | 25 | 27 | 0 | 0
Stage II FAS for Persistence | 0 | 0 | 24 | 28 | 0 | 0
Safety Analysis Set | 0 | 0 | 27 (Two participants were incorrectly assessed by Investigator as having received MenACYW Conjugate vaccine in study MET49 and underwent randomization to Group 4 instead of Group 3. These participants were included in Group 3 for safety analysis as per actual vaccination received.) | 25 | 0 | 0
Completed | 0 | 0 | 25 | 26 | 0 | 0
Not Completed | 0 | 0 | 6 | 13 | 0 | 0
Not completed — Non-compliance with the protocol | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 5 | 9 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all enrolled participants.
Groups:
- Group 1: MenACYW Conjugate Vaccine (MET 49 - Menomune-primed Participants): Participants who received a single dose of Menomune vaccine in a previous study MET49, provided a blood sample for assessment of antibody persistence (at enrollment [Day 0]) followed by a single IM dose of MenACYW Conjugate vaccine, at Day 0, during Stage I in the present study (MEQ00066).
- Group 4: MenACYW Conjugate Vaccine (MET49: MenACYW-primed Participants): Participants who received a single dose of MenACYW Conjugate vaccine in a previous study MET49, provided a blood sample for assessment of antibody persistence at enrollment (Day 0), during Stage I in the present study (MEQ00066), followed by receiving a single IM dose of MenACYW Conjugate vaccine at Stage II in the present study (MEQ00066).
- Total: Total of all reporting groups
Arm/Group | Group 1: MenACYW Conjugate Vaccine (MET 49 - Menomune-primed Participants) | Group 2: MenACYW Conjugate Vaccine (MET49 - MenACYW Conjugate Vaccine-primed Participants) | Group 3: MenACYW Conjugate Vaccine (MET49: Menomune-primed Participants) | Group 4: MenACYW Conjugate Vaccine (MET49: MenACYW-primed Participants) | Group 5: Menomune-primed Participants (MET44) | Group 6: MenACYW Conjugate Vaccine-primed Participants (MET44) | Total
Number analyzed (Participants) | 139 | 176 | 31 | 39 | 26 | 60 | 471
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.6 (7.48) | 69.8 (7.43) | 69.2 (7.14) | 69.7 (6.39) | 70.5 (5.69) | 71.4 (6.28) | 70.2 (7.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 111 | 15 | 27 | 11 | 42 | 291
  Male | 54 | 65 | 16 | 12 | 15 | 18 | 180
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 127 | 158 | 27 | 32 | 25 | 57 | 426
  Asian | 0 | 2 | 0 | 0 | 0 | 0 | 2
  Black or African American | 11 | 16 | 3 | 7 | 0 | 3 | 40
  Native American or Alaska Native | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Mixed Origin | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Stage I: Percentage of Participants With Seroresponse for Meningococcal Serogroups A, C, W & Y Measured by Serum Bactericidal Assay Using Human Complement (hSBA) After Vaccination With MenACYW Conjugate Vaccine in Study MEQ00066: Group 1 (Menomune-primed)
Description: Antibody titers against meningococcal serogroups A, C, W, and Y were measured by hSBA. The hSBA vaccine seroresponse was defined as a post-vaccination hSBA titer greater than or equal to (>=) 1:16 for participants with pre-vaccination hSBA titer less than (<) 1:8, or a >= 4-fold increase in hSBA titer from pre-vaccination to post-vaccination for participants with pre-vaccination hSBA titer >= 1:8.
Time Frame: Day 30 (post-vaccination) in study MEQ00066
Population: Stage I Day 30 Per-Protocol Analysis Set (PPAS) population: participants of Groups 1 and 2 who received 1 dose of vaccine in MEQ00066 and had valid serology result for at least 1 serogroup from a blood sample provided 30 days (+14) post-vaccination with no relevant protocol deviations. 'Number analyzed'=participants with available data for each specified category. For this outcome measure, data were not planned to be collected and analyzed for Groups 3, 4, 5 and 6 as pre-specified in protocol.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine (MET 49 - Menomune-primed Participants)
Number analyzed (Participants) | 130
percentage of participants
  Serogroup A | 60.8 [51.8 to 69.2]
  Serogroup C: number analyzed (Participants) | 129
  Serogroup C | 55.0 [46.0 to 63.8]
  Serogroup W | 49.2 [40.4 to 58.1]
  Serogroup Y | 49.2 [40.4 to 58.1]

2. Secondary Outcome: Stage I: Percentage of Participants With Vaccine Seroresponse for Meningococcal Serogroups A, C, W, and Y Measured by hSBA After Vaccination With MenACYW Conjugate Vaccine in Study MEQ00066: Group 2 (MenACYW Conjugate Vaccine-primed Participants)
Description: Antibody titers against meningococcal serogroups A, C, W, and Y were measured by hSBA. The hSBA vaccine seroresponse was defined as a post-vaccination hSBA titer >= 1:16 for participants with pre-vaccination hSBA titer < 1:8, or a >= 4-fold increase in hSBA titer from pre-vaccination to post-vaccination for participants with pre-vaccination hSBA titer >= 1:8.
Time Frame: Day 30 (post-vaccination) in study MEQ00066
Population: Analysis was performed on Stage I Day 30 PPAS population. For this outcome measure, data were not planned to be collected and analyzed for Groups 3, 4, 5 and 6 as pre-specified in the protocol.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 2: MenACYW Conjugate Vaccine (MET49 - MenACYW Conjugate Vaccine-primed Participants)
Number analyzed (Participants) | 145
percentage of participants
  Serogroup A | 79.3 [71.8 to 85.6]
  Serogroup C | 93.1 [87.7 to 96.6]
  Serogroup W | 90.3 [84.3 to 94.6]
  Serogroup Y | 92.4 [86.8 to 96.2]

3. Secondary Outcome: Stage I: Percentage of Participants With Vaccine Seroresponse for Meningococcal Serogroups A, C, W, and Y Measured by hSBA at Day 6 After Vaccination With MenACYW Conjugate Vaccine in Study MEQ00066: Groups 1 and 2
Description: as for outcome 2
Time Frame: Day 6 (post-vaccination) in study MEQ00066
Population: Analysis was performed on Stage I Day 6 PPAS which included participants of Groups 1 and 2 who had received the study MEQ00066 vaccine and had a valid serology result for at least 1 serogroup from a blood sample provided 6 days (window, 5 to 7) post-vaccination with no relevant protocol deviations. For this outcome measure, data were not planned to be collected and analyzed for Groups 3, 4, 5 and 6 as pre-specified in the protocol.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine (MET 49 - Menomune-primed Participants) | Group 2: MenACYW Conjugate Vaccine (MET49 - MenACYW Conjugate Vaccine-primed Participants)
Number analyzed (Participants) | 62 | 58
percentage of participants
  Serogroup A | 8.1 [2.7 to 17.8] | 36.2 [24.0 to 49.9]
  Serogroup C | 8.1 [2.7 to 17.8] | 77.6 [64.7 to 87.5]
  Serogroup W | 6.5 [1.8 to 15.7] | 70.7 [57.3 to 81.9]
  Serogroup Y | 8.1 [2.7 to 17.8] | 72.4 [59.1 to 83.3]

4. Secondary Outcome: Stage I: Geometric Mean Titers (GMTs) of Antibodies Against Meningococcal Serogroups A, C, W, and Y Measured by hSBA Before and After Vaccination With MenACYW Conjugate Vaccine in Study MEQ00066 (Groups 1 to 4)
Description: GMTs of antibodies against meningococcal serogroups A, C, W, and Y 135 were measured by hSBA. Titers are expressed in terms of 1/dilution. At Baseline, Group 1 was equivalent to Group 3 (both groups were Menomune-primed in MET49) and Group 2 was equivalent to Group 4 (both groups were MenACYW Conjugate Vaccine-primed in MET49), therefore it was planned to collect and present pooled data of Groups 1 and 3 and Groups 2 and 4 for Day 0 (pre-vaccination) in this outcome measure. Here, "0" in the number analyzed field for Day 30 signifies that data were not planned to be collected and analyzed for Groups 3 and 4 participants as pre-specified in the protocol.
Time Frame: Day 0 (pre-vaccination) and Day 30 (post-vaccination) in study MEQ00066
Population: Analysis was performed on the Stage I Full Analysis Set (FAS) population for persistence which included Groups 1, 2, 3, 4, 5 and 6 participants who had a valid serology result for at least 1 serogroup from a pre-vaccination blood sample. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Groups:
- Pooled Groups 1 and 3: MenACYW Conjugate Vaccine (MET49: Menomune-primed Participants): Included all participants of Groups 1 and 3 who received a single dose of Menomune vaccine in a previous study MET49. Participants in each group provided a blood sample for assessment of antibody persistence at enrollment (Day 0) in the present study (MEQ00066). In addition, Group 1 participants received a single IM dose of MenACYW Conjugate vaccine at Day 0 in the present study (MEQ00066).
- Pooled Groups 2 and 4: MenACYW Conjugate Vaccine (MET49: MenACYW-primed Participants): Included all participants of Groups 2 and 4 who received a single dose of MenACYW Conjugate vaccine in a previous study MET49. Participants in each group provided a blood sample for assessment of antibody persistence at enrollment (Day 0) in the present study (MEQ00066). In addition, Group 2 participants received a single IM dose of MenACYW Conjugate vaccine at Day 0 in the present study (MEQ00066).
Arm/Group | Group 1: MenACYW Conjugate Vaccine (MET 49 - Menomune-primed Participants) | Group 2: MenACYW Conjugate Vaccine (MET49 - MenACYW Conjugate Vaccine-primed Participants) | Pooled Groups 1 and 3: MenACYW Conjugate Vaccine (MET49: Menomune-primed Participants) | Pooled Groups 2 and 4: MenACYW Conjugate Vaccine (MET49: MenACYW-primed Participants)
Number analyzed (Participants) | 138 | 175 | 169 | 214
titers
  Serogroup A: Day 0 (pre-vaccination) | 11.6 [9.40 to 14.3] | 11.8 [9.77 to 14.4] | 11.6 [9.53 to 14.1] | 12.2 [10.2 to 14.6]
  Serogroup A: Day 30 (post-vaccination): number analyzed (Participants) | 138 | 174 | 0 | 0
  Serogroup A: Day 30 (post-vaccination) | 57.6 [42.8 to 77.6] | 144 [110 to 188] |  |
  Serogroup C: Day 0 (pre-vaccination) | 8.85 [6.87 to 11.4] | 17.7 [14.0 to 22.5] | 8.47 [6.76 to 10.6] | 17.7 [14.3 to 21.9]
  Serogroup C: Day 30 (post-vaccination): number analyzed (Participants) | 137 | 174 | 0 | 0
  Serogroup C: Day 30 (post-vaccination) | 56.7 [40.7 to 78.9] | 568 [447 to 721] |  |
  Serogroup W: Day 0 (pre-vaccination) | 6.68 [5.24 to 8.50] | 14.5 [11.5 to 18.3] | 6.54 [5.28 to 8.11] | 14.2 [11.6 to 17.4]
  Serogroup W: Day 30 (post-vaccination): number analyzed (Participants) | 138 | 174 | 0 | 0
  Serogroup W: Day 30 (post-vaccination) | 31.5 [23.1 to 42.9] | 377 [290 to 490] |  |
  Serogroup Y: Day 0 (pre-vaccination) | 8.08 [5.91 to 11.0] | 15.5 [12.2 to 19.7] | 7.49 [5.72 to 9.82] | 15.3 [12.3 to 19.1]
  Serogroup Y: Day 30 (post-vaccination): number analyzed (Participants) | 138 | 174 | 0 | 0
  Serogroup Y: Day 30 (post-vaccination) | 41.8 [30.2 to 57.7] | 478 [371 to 617] |  |

5. Secondary Outcome: Stage I: Geometric Mean Titers of Antibodies Against Meningococcal Serogroups A, C, W, and Y Measured by hSBA: Groups 5 and 6
Description: GMTs of antibodies against meningococcal serogroups A, C, W, and Y were measured by hSBA. Titers were expressed in terms of 1/dilution.
Time Frame: Day 0 (pre-vaccination in MEQ00066)
Population: Analysis was performed on Stage I FAS population.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Groups:
- Group 5: Menomune-primed Participants (MET44): Participants who received a single dose of Menomune vaccine in a previous study MET44, provided a blood sample for assessment of antibody persistence at enrollment (Day 0, Stage I) in the present study (MEQ00066). These participants did not receive any vaccination in the present study (MEQ00066).
- Group 6: MenACYW Conjugate Vaccine-primed Participants (MET44): Participants who received a single dose of MenACYW Conjugate vaccine in a previous study MET44, provided a blood sample for assessment of antibody persistence at enrollment (Day 0, Stage I) in the present study (MEQ00066). These participants did not receive any vaccination in the present study (MEQ00066).
Arm/Group | Group 5: Menomune-primed Participants (MET44) | Group 6: MenACYW Conjugate Vaccine-primed Participants (MET44)
Number analyzed (Participants) | 26 | 59
titers
  Serogroup A | 9.64 [5.18 to 17.9] | 9.00 [6.44 to 12.6]
  Serogroup C | 7.58 [4.11 to 14.0] | 11.9 [7.67 to 18.5]
  Serogroup W | 4.95 [3.39 to 7.22] | 11.9 [7.97 to 17.8]
  Serogroup Y | 7.19 [4.09 to 12.6] | 11.2 [7.24 to 17.5]

6. Secondary Outcome: Stage I: Percentage of Participants With Antibody Titers >=1:4 and >=1:8 Against Meningococcal Serogroups A, C, W, and Y Measured by hSBA After Primary Vaccination With Menomune Vaccine or MenACYW Conjugate Vaccine: Groups 1 to 6
Description: Antibody titers against meningococcal serogroups A, C, W, and Y were measured by hSBA.
Time Frame: Day 0 (pre-vaccination) in study MEQ00066
Population: Analysis was performed on Stage I FAS population. At Baseline, Group 1 was equivalent to Group 3 (both groups were Menomune-primed in MET49) and Group 2 was equivalent to Group 4 (both groups were MenACYW Conjugate Vaccine-primed in MET49), therefore it was planned to collect and present pooled data of Groups 1 and 3 and Groups 2 and 4 for Day 0 (pre-vaccination) in this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine (MET 49 - Menomune-primed Participants) | Group 2: MenACYW Conjugate Vaccine (MET49 - MenACYW Conjugate Vaccine-primed Participants) | Pooled Groups 1 and 3: MenACYW Conjugate Vaccine (MET49: Menomune-primed Participants) | Pooled Groups 2 and 4: MenACYW Conjugate Vaccine (MET49: MenACYW-primed Participants) | Group 5: Menomune-primed Participants (MET44) | Group 6: MenACYW Conjugate Vaccine-primed Participants (MET44)
Number analyzed (Participants) | 138 | 175 | 169 | 214 | 26 | 59
percentage of participants
  Serogroup A: >= 1:4 | 86.2 [79.3 to 91.5] | 89.1 [83.6 to 93.3] | 85.8 [79.6 to 90.7] | 87.9 [82.7 to 91.9] | 84.6 [65.1 to 95.6] | 81.4 [69.1 to 90.3]
  Serogroup A: >= 1:8 | 65.2 [56.6 to 73.1] | 65.1 [57.6 to 72.2] | 65.7 [58.0 to 72.8] | 65.0 [58.2 to 71.3] | 50.0 [29.9 to 70.1] | 55.9 [42.4 to 68.8]
  Serogroup C: >= 1:4 | 71.0 [62.7 to 78.4] | 89.1 [83.6 to 93.3] | 69.8 [62.3 to 76.6] | 89.7 [84.8 to 93.4] | 73.1 [52.2 to 88.4] | 79.7 [67.2 to 89.0]
  Serogroup C: >= 1:8 | 49.3 [40.7 to 57.9] | 74.3 [67.1 to 80.6] | 47.9 [40.2 to 55.7] | 73.4 [66.9 to 79.2] | 42.3 [23.4 to 63.1] | 59.3 [45.7 to 71.9]
  Serogroup W: >= 1:4 | 64.5 [55.9 to 72.4] | 81.1 [74.5 to 86.6] | 64.5 [56.8 to 71.7] | 83.2 [77.5 to 87.9] | 61.5 [40.6 to 79.8] | 79.7 [67.2 to 89.0]
  Serogroup W: >= 1:8 | 40.6 [32.3 to 49.3] | 66.9 [59.4 to 73.8] | 39.6 [32.2 to 47.4] | 66.8 [60.1 to 73.1] | 38.5 [20.2 to 59.4] | 66.1 [52.6 to 77.9]
  Serogroup Y: >= 1:4 | 53.6 [44.9 to 62.1] | 81.1 [74.5 to 86.6] | 53.3 [45.4 to 61.0] | 79.4 [73.4 to 84.6] | 57.7 [36.9 to 76.6] | 71.2 [57.9 to 82.2]
  Serogroup Y: >= 1:8 | 42.0 [33.7 to 50.7] | 69.1 [61.7 to 75.9] | 40.8 [33.3 to 48.6] | 68.2 [61.5 to 74.4] | 46.2 [26.6 to 66.6] | 59.3 [45.7 to 71.9]

7. Secondary Outcome: Stage II: Geometric Mean Titers of Antibodies Against Meningococcal Serogroups A, C, W, and Y Measured by hSBA After Primary Vaccination With Menomune Vaccine or MenACYW Conjugate Vaccine: Groups 3 and 4
Description: as for outcome 5
Time Frame: 5 years post primary vaccination (with Menomune or MenACYW Conjugate vaccine) in study MET49
Population: Analysis was performed on Stage II FAS for persistence that included participants in Groups 3 and 4 who had a valid serology result for at least 1 serogroup from pre-vaccination blood sample (5-year antibody persistence). Data for this outcome measure was not planned to be collected and analyzed for Groups 1, 2, 5 and 6 as pre-specified in the protocol.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 3: MenACYW Conjugate Vaccine (MET49: Menomune-primed Participants) | Group 4: MenACYW Conjugate Vaccine (MET49: MenACYW-primed Participants)
Number analyzed (Participants) | 24 | 28
titers
  Serogroup A | 8.72 [5.42 to 14.0] | 15.6 [9.48 to 25.7]
  Serogroup C | 3.78 [2.59 to 5.50] | 7.25 [3.68 to 14.3]
  Serogroup W | 4.62 [2.50 to 8.56] | 7.07 [4.17 to 12.0]
  Serogroup Y | 4.00 [2.35 to 6.81] | 5.25 [3.32 to 8.31]

8. Secondary Outcome: Stage II: Geometric Mean Titers of Antibodies Against Meningococcal Serogroups A, C, W, and Y Measured by rSBA After Primary Vaccination With Menomune Vaccine or MenACYW Conjugate Vaccine: Groups 3 and 4
Description: GMTs of antibodies against meningococcal serogroups A, C, W, and Y were measured by rSBA. Titers were expressed in terms of 1/dilution.
Time Frame: 5 years post primary vaccination (with Menomune or MenACYW Conjugate vaccine) in study MET49
Population: Analysis was performed on Stage II FAS for persistence. Data for this outcome measure was not planned to be collected and analyzed for Groups 1, 2, 5 and 6 as pre-specified in the protocol.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 3: MenACYW Conjugate Vaccine (MET49: Menomune-primed Participants) | Group 4: MenACYW Conjugate Vaccine (MET49: MenACYW-primed Participants)
Number analyzed (Participants) | 24 | 28
titers
  Serogroup A | 24.0 [6.93 to 83.0] | 40.0 [12.4 to 129]
  Serogroup C | 13.8 [5.16 to 37.2] | 64.0 [24.7 to 166]
  Serogroup W | 9.79 [3.37 to 28.4] | 25.0 [8.48 to 73.6]
  Serogroup Y | 4.00 [1.84 to 8.70] | 34.5 [10.9 to 109]

9. Secondary Outcome: Stage II: Percentage of Participants With Antibody Titers >=1:4 and >=1:8 Against Meningococcal Serogroups A, C, Y, and W Measured by hSBA After Primary Vaccination With Menomune Vaccine or MenACYW Conjugate Vaccine: Groups 3 and 4
Description: Antibody titers against meningococcal serogroups A, C, W, and Y were measured by hSBA.
Time Frame: 5 years post primary vaccination (with Menomune or MenACYW Conjugate vaccine) in study MET49
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 3: MenACYW Conjugate Vaccine (MET49: Menomune-primed Participants) | Group 4: MenACYW Conjugate Vaccine (MET49: MenACYW-primed Participants)
Number analyzed (Participants) | 24 | 28
percentage of participants
  Serogroup A: >= 1:4 | 79.2 [57.8 to 92.9] | 89.3 [71.8 to 97.7]
  Serogroup A: >= 1:8 | 58.3 [36.6 to 77.9] | 78.6 [59.0 to 91.7]
  Serogroup C: >= 1:4 | 50.0 [29.1 to 70.9] | 64.3 [44.1 to 81.4]
  Serogroup C: >= 1:8 | 20.8 [7.1 to 42.2] | 28.6 [13.2 to 48.7]
  Serogroup W: >= 1:4 | 33.3 [15.6 to 55.3] | 64.3 [44.1 to 81.4]
  Serogroup W: >= 1:8 | 29.2 [12.6 to 51.1] | 46.4 [27.5 to 66.1]
  Serogroup Y: >= 1:4 | 37.5 [18.8 to 59.4] | 50.0 [30.6 to 69.4]
  Serogroup Y: >= 1:8 | 29.2 [12.6 to 51.1] | 42.9 [24.5 to 62.8]

10. Secondary Outcome: Stage II: Percentage of Participants With Antibody Titers >=1:8 and >=1:128 Against Meningococcal Serogroups A, C, Y, and W Measured by rSBA After Primary Vaccination With Menomune Vaccine or MenACYW Conjugate Vaccine: Groups 3 and 4
Description: Antibody titers against meningococcal serogroups A, C, W, and Y were measured by rSBA.
Time Frame: 5 years post primary vaccination (with Menomune or MenACYW Conjugate vaccine) in study MET49
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 3: MenACYW Conjugate Vaccine (MET49: Menomune-primed Participants) | Group 4: MenACYW Conjugate Vaccine (MET49: MenACYW-primed Participants)
Number analyzed (Participants) | 24 | 28
percentage of participants
  Serogroup A: >= 1:8 | 45.8 [25.6 to 67.2] | 53.6 [33.9 to 72.5]
  Serogroup A: >= 1:128 | 41.7 [22.1 to 63.4] | 50.0 [30.6 to 69.4]
  Serogroup C: >= 1:8 | 45.8 [25.6 to 67.2] | 75.0 [55.1 to 89.3]
  Serogroup C: >= 1:128 | 25.0 [9.8 to 46.7] | 53.6 [33.9 to 72.5]
  Serogroup W: >= 1:8 | 29.2 [12.6 to 51.1] | 50.0 [30.6 to 69.4]
  Serogroup W: >= 1:128 | 29.2 [12.6 to 51.1] | 46.4 [27.5 to 66.1]
  Serogroup Y: >= 1:8 | 12.5 [2.7 to 32.4] | 50.0 [30.6 to 69.4]
  Serogroup Y: >= 1:128 | 12.5 [2.7 to 32.4] | 50.0 [30.6 to 69.4]

ADVERSE EVENTS:
Time Frame: Unsolicited adverse event (AE) data were collected from Day 0 (pre-vaccination) up to Day 30 (post-vaccination). The solicited reactions (SR) were collected within 7 days post-vaccination. Serious AEs data were collected throughout the study (i.e., up to 30 days post-vaccination for Groups 1 and 2; and 2 years post-vaccination for Groups 3 and 4 in the current study)
Description: Analysis performed on SafAS population. Safety data were planned to be collected and reported for participants revaccinated with MenACYW conjugate vaccine (i.e., participants in Groups 1 and 2 during Stage I, and participants in Groups 3 and 4 during Stage II). Since participants in Groups 5 and 6 were not vaccinated in MEQ00066 as pre-specified in the protocol, safety data were not planned to be collected and reported for Groups 5 and 6.
Groups:
- Stage I - Group 1: MenACYW Conjugate Vaccine (MET 49 - Menomune-primed Participants): Participants who received a single dose of Menomune vaccine in a previous study MET49, provided a blood sample for assessment of antibody persistence (at enrollment [Day 0]) followed by a single IM dose of MenACYW Conjugate vaccine, at Day 0, during Stage I in the present study (MEQ00066).
- Stage I - Group 2: MenACYW Conjugate Vaccine (MET49 - MenACYW Conjugate Vaccine-primed Participants): Participants who received a single dose of MenACYW Conjugate vaccine in a previous study MET49, provided a blood sample for assessment of antibody persistence (at enrollment [Day 0]) followed by a single IM dose of MenACYW Conjugate vaccine at Day 0, during Stage I in the present study (MEQ00066).
- Stage II - Group 3: MenACYW Conjugate Vaccine (MET49: Menomune-primed Participants): Participants who received a single dose of Menomune vaccine in a previous study MET49, provided a blood sample for assessment of antibody persistence at enrollment (Day 0) during Stage I in the present study (MEQ00066), followed by receiving a single IM dose of MenACYW Conjugate vaccine at Stage II in the present study (MEQ00066).
- Stage II - Group 4: MenACYW Conjugate Vaccine (MET49: MenACYW-primed Participants): Participants who received a single dose of MenACYW Conjugate vaccine in a previous study MET49, provided a blood sample for assessment of antibody persistence at enrollment (Day 0, Stage I) in the present study (MEQ00066), followed by receiving a single IM dose of MenACYW Conjugate vaccine at Stage II in the present study (MEQ00066).
Arm/Group | Stage I - Group 1: MenACYW Conjugate Vaccine (MET 49 - Menomune-primed Participants) | Stage I - Group 2: MenACYW Conjugate Vaccine (MET49 - MenACYW Conjugate Vaccine-primed Participants) | Stage II - Group 3: MenACYW Conjugate Vaccine (MET49: Menomune-primed Participants) | Stage II - Group 4: MenACYW Conjugate Vaccine (MET49: MenACYW-primed Participants)
All-Cause Mortality (participants affected / at risk) | 0/151 | 0/162 | 0/27 | 0/25
Serious Adverse Events (participants affected / at risk) | 2/151 | 1/162 | 0/27 | 1/25
Other Adverse Events (participants affected / at risk) | 55/151 | 62/162 | 10/27 | 5/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage I - Group 1: MenACYW Conjugate Vaccine (MET 49 - Menomune-primed Participants) (N=151) | Stage I - Group 2: MenACYW Conjugate Vaccine (MET49 - MenACYW Conjugate Vaccine-primed Participants) (N=162) | Stage II - Group 3: MenACYW Conjugate Vaccine (MET49: Menomune-primed Participants) (N=27) | Stage II - Group 4: MenACYW Conjugate Vaccine (MET49: MenACYW-primed Participants) (N=25)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epithelioid Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage I - Group 1: MenACYW Conjugate Vaccine (MET 49 - Menomune-primed Participants) (N=151) | Stage I - Group 2: MenACYW Conjugate Vaccine (MET49 - MenACYW Conjugate Vaccine-primed Participants) (N=162) | Stage II - Group 3: MenACYW Conjugate Vaccine (MET49: Menomune-primed Participants) (N=27) | Stage II - Group 4: MenACYW Conjugate Vaccine (MET49: MenACYW-primed Participants) (N=25)
Injection Site Erythema (General disorders) | 11 (11) | 6 (6) | 2 (2) | 1 (1)
Injection Site Pain (General disorders) | 32 (33) | 27 (27) | 6 (6) | 3 (3)
Malaise (General disorders) | 22 (22) | 22 (22) | 4 (4) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 30 (30) | 35 (35) | 5 (5) | 4 (4)
Headache (Nervous system disorders) | 21 (21) | 30 (31) | 5 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable participant matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2020-09-11): https://cdn.clinicaltrials.gov/large-docs/42/NCT04142242/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-30): https://cdn.clinicaltrials.gov/large-docs/42/NCT04142242/SAP_001.pdf